CLINICAL TRIAL: NCT07345208
Title: An Open Label, Randomized Non-Inferiority Trial Comparing Safety and Immunogenicity of Intradermal Versus Intramuscular Administration of Registered Rabies Vaccine (by Popular Pharmaceuticals PLC.) in Healthy Bangladeshi Population
Brief Title: Safety and Immunogenicity of ID vs IM Rabies Vaccine
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Popular Pharmaceuticals PLC. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR-25035
Record Dates: First submitted 2025-12-03; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rabies
Keywords: pre-exposure prophylaxis; intradermal; rabies vaccine; clinical trial; intramuscular; safety; immunogenicity; non-inferiority
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: Since we already have an established intramuscular vaccine regimen for Rabies, we have chosen to follow a randomized, single-blinded, non-inferiority trial to assess the immunogenicity of the intradermal Rabies vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm-1 (Experimental): 0.2 ml (0.1 ml in both deltoid regions) Inj. Rabivax ID/SC via the intradermal (ID) route
  Interventions: Biological: Rabies vaccine
- Reference Arm-2 (Active Comparator): 1 ml (in the deltoid region of one arm) inj. Rabivax IM via the intramuscular (IM) route.
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: Rabies vaccine — The intradermal rabies vaccine is designed to elicit an immune response in the skin. The skin is composed of three layers, from outermost to innermost: the epidermis, dermis, and hypodermis, where the dermis is further divided into two sub-layers: the superficial papillary dermis and the deeper reticular dermis. The papillary dermis is 100-300 μm thick and is the target layer for ID immunization. This layer is rich in antigenpresenting cells (APCs), including dermal dendritic cells (DDCs) and Langerhans cells. DDCs capture antigens in the dermis and migrate to the regional lymph nodes, which present antigens to T-cells, triggering their activation. Soluble antigens also migrate to lymph nodes, leading to the activation of B-cells. Because of the high concentration of APCs in the dermis, ID delivery of reduced antigen doses (typically 20% to 30% of the standard amount) can elicit immune responses comparable to those achieved with standard doses administered intramuscularly.
  Other Names: inj. Rabivax ID/SC
  Arms: Test Arm-1
Biological: Rabies vaccine — Rabies vaccine is an active immunizing agent used to prevent infection caused by the rabies virus. The vaccine works by causing the body to produce its own protection (antibodies) against the rabies virus.
  Other Names: Inj. Rabivax IM
  Arms: Reference Arm-2

SUMMARY:
Background:

Burden: Rabies is a viral zoonotic disease that is 100% fatal if left untreated. Globally, Bangladesh is ranked third in terms of rabies infections. In 2009, the estimated human fatality from rabies in Bangladesh surpassed 2,000. However, the death toll has steadily declined to 26 in 2020, owing to the implementation of the 'National Rabies Elimination Program' beginning in 2010, which included the introduction of the cell culture vaccine. Though this infection is entirely preventable by vaccination, the available intramuscular regimen is costly and requires multiple high doses.

Knowledge gap: The safety and immunogenicity of an intradermal rabies vaccine regimen in the Bangladeshi population needs to be assessed to comply with the recommendation of DGDA to obtain approval to be administered through an alternate route.

Relevance: Intradermal rabies vaccine administration is a safe method that reduces the amount of vaccine needed and the number of doses required by producing immunogenicity similar to that of the intramuscular regimen. This translates to 60-80% cost reductions while preserving the safety and immunogenicity of the vaccine. The intramuscular rabies vaccine by Popular Pharmaceuticals PLC has already been granted marketing authorization by DGDA. However, the vaccine's administration via the intradermal route is yet to receive approval from DGDA for marketing as per the regulatory requirements.

Hypothesis: The immunogenicity and safety of the Intradermal rabies vaccine (Popular Pharmaceutical PLC) will be non-inferior to the intramuscular regimen of the same vaccine.

Objectives:

1. To compare the seroconversion level of the intradermal rabies vaccine to the intramuscular regimen by Popular Pharmaceuticals PLC. in healthy Bangladeshi individuals
2. To compare the safety of the intradermal rabies vaccine to the intramuscular regimen by Popular Pharmaceuticals PLC. in healthy Bangladeshi individuals

Methods: This will be an open-label, non-inferiority, single-blinded, randomized controlled trial where the safety and immunogenicity of the intradermal rabies vaccine will be assessed compared with the standard intramuscular regimen, both by Popular Pharmaceuticals PLC., amongst healthy individuals. The study will be conducted at the Infectious Disease and Tropical Medicine Department (Surya Kanta Hospital), Mymensingh Medical College Hospital, Mymensingh. We will enroll 90 participants and randomly assign them to two equal groups: a test group and a reference group. The test groups will receive 0.2 ml Inj. Rabivax intradermally (0.1 ml in each arm), whereas the reference group will receive 1 ml Injectable Rabivax (2.5 IU/ml) intramuscularly. The participants will be followed up on days 21, 35, and 187 for clinical and biochemical evaluation. A comparative analysis of safety and immunogenicity will be conducted on intradermal and intramuscular administration based on the collected data.

Outcome measures/variables:

* A seroconversion level of 0.5 IU/ml or more when tested for Rabies Virus Neutralizing Antibody (RVNA) following intradermal vaccination by Popular Pharmaceuticals PLC. during the study period
* Non-inferior safety parameters of the intradermal rabies vaccine regimen in comparison with the available intramuscular regimen by Popular Pharmaceuticals PLC.

DETAILED DESCRIPTION:
Epidemiology of Rabies:

Rabies is a vaccine-preventable zoonotic viral disease that primarily targets the central nervous system, leading to severe neurological symptoms and, if untreated, is 100% fatal. It is transmitted through the bite or saliva of an infected animal, with dogs being the most common source of human infections worldwide. The virus travels from the site of infection through the peripheral nerves to the brain, where it causes encephalitis, characterized by confusion, agitation, paralysis, and ultimately, coma and death.

Globally, rabies is responsible for around 59,000 deaths each year, with the majority occurring in Asia and Africa. An alarming 40% of those affected are children under the age of 15. This infection comes with an economic burden of $8.6 billion annually. A similar scenario prevails in Bangladesh. Bangladesh is ranked third globally in terms of rabies infections, right after China and India. In 2009, rabies-related human deaths in Bangladesh were estimated to exceed 2,000. However, the death toll has steadily declined to 26 in 2020, owing to the implementation of the 'National Rabies Elimination Program' beginning in 2010, which included the introduction of the cell culture vaccine.

Treatment of Rabies from a Bangladeshi Perspective:

Despite being ultimately fatal when symptoms show, rabies is 100% preventable by vaccination. Louis Pasteur was the first to administer the rabies vaccine to a patient in 1885. Currently, two types of vaccines are available for protection against rabies: nerve tissue vaccines and cell culture vaccines. The World Health Organization (WHO) recommends replacing nerve tissue vaccines with more effective and safer cell culture-based vaccines as soon as possible. Recent advancements in cell culture vaccines have made them more affordable and require smaller doses. Cell-culture-based rabies vaccines can be administered through two different routes: intramuscular (IM) and intradermal (ID). As per the National Guideline for Animal Bite Management in Bangladesh, (i) a 1-site IM regimen or 2-site ID regimen for Pre-exposure Prophylaxis (PrEP), and (ii) a 1-site IM regimen or 2-site ID regimen for Post-exposure Prophylaxis (PEP) is available for Rabies prevention. The IM regimen is more commonly used in clinical settings, as observed in various studies. However, the IM regimen has been found to elicit a serious adverse event (SAE) in a previous study. Seven days after receiving an intramuscular rabies vaccine regimen, Bell's Palsy was reported as a suspected unexpected SAE. Moreover, multiple studies conducted worldwide have demonstrated the superiority of the ID regimen over IM in terms of seroprotection.

The introduction of an intradermal rabies vaccine regimen in Bangladesh could have significant public health implications. As a low-resource country with a high burden of rabies, Bangladesh could benefit greatly from a more cost-effective vaccination method. Given that the intradermal route uses significantly less vaccine (up to 80% less per dose) and reduces costs by about 75% compared to intramuscular injection, its adoption could lead to much wider vaccine coverage within budgetary limits and a substantial decrease in the economic burden of rabies. This could potentially lead to increased accessibility of rabies prevention, especially in rural and underserved areas where cost is a major barrier to vaccination. Furthermore, the dose-sparing nature of the intradermal route could help mitigate vaccine shortages, which are occasionally reported worldwide. By conducting this trial, we aim to provide local evidence to support the adoption of this WHO-recommended approach, potentially revolutionizing rabies prevention strategies in Bangladesh.

This study seeks to determine the safety and immunogenicity of intradermally administered Inj. Rabivax ID/SC by Popular Pharmaceuticals PLC. (Test) and Inj. Rabivax IM (2.5 IU/ml) by the same manufacturer (Reference) in healthy participants in pre-exposure prophylactic doses.

What is seroconversion? The production of antibodies in an individual following vaccination or exposure to any antigen is called seroconversion. According to WHO, an adequate antibody response is usually defined as 0.5 IU/ml or more at 14 and 28-30 days following the final vaccination dose. The Advisory Committee on Immunization Practices (ACIP) has endorsed this Rabies Virus Neutralizing Antibody (RVNA) level, thereby replacing the previously established minimum acceptable rabies antibody titer of 0.1-0.3 IU/ml (16). This higher limit offers a more conservative approach to determining inadequate response and booster requirements. RVNA level is usually assessed using one of the two serological assays: rapid fluorescent focus inhibition test (RFFIT) or fluorescent antibody virus neutralization (FAVN). In this study, we will focus on the RFFIT for the assessment of RVNA level. RFFIT is a serological assay that quantifies the neutralizing capacity of rabies-specific antibodies, reflecting their ability to inhibit viral infection of susceptible cells. This investigational procedure utilizes serial fivefold dilutions of patient serum, which are subsequently combined with a standardized challenge dose of live rabies virus. Following incubation, the serum/virus mixtures are introduced to susceptible cell cultures. The presence of RVNA is determined by assessing the inhibition of viral cytopathic effect through fluorescent antibody staining. The endpoint titer is calculated based on the highest serum dilution that demonstrates significant neutralization. Since the World Health Organization (WHO) and the Advisory Committee on Immunization Practices (ACIP) consider an RVNA level of complete neutralization at a 1:5 serum dilution by the RFFIT test as proof of a sufficient immune response to rabies vaccination, this test will provide us with the accurate immunogenicity of the test vaccine.

The assessment of the seroconversion rate among the enrolled participants will be one of the primary outcome measures of this study. The seroconversion rate is defined as the proportion of subjects with RVNA level ≥0.5 IU/mL, measured 4 weeks after vaccination completion. We will perform a comparative analysis to determine the non-inferiority of seroconversion rates between participants receiving intradermal and intramuscular rabies vaccinations.

Safety Profile Rabies vaccine production involves three principal types: the now largely obsolete nerve tissue vaccines, contemporary cell culture vaccines, and vaccines derived from embryonated eggs. WHO guidelines endorse cell culture and embryonated egg rabies vaccines over nerve tissue vaccines since the latter pose risks of severe adverse events and reduced immunogenicity, including the potential for rabies transmission due to incomplete virus inactivation. In comparison, cell culture and embryonated egg vaccines exhibit a favorable safety profile and are generally well-tolerated. In our study, we will use purified Vero cell vaccine (PVRV) for both the test and reference groups. By utilizing a serum-free medium and an animal-origin-free trypsin-like enzyme, this cell culture vaccine is designed to minimize the risk of hypersensitivity and the transmission of contaminants, including bacteria, fungi, and mycoplasma. Furthermore, Frazatti-Gallina et al. demonstrated the safety of PVRV in mouse models. A Chinese trial by the manufacturers of our study vaccines established the safety of this vaccine in murine models. In addition, the vaccine has proved to be safe in healthy participants of different age groups. The safety of these rabies vaccines in pregnant women has also been demonstrated in prior studies. These purified Vero cell vaccines produce mild to moderate adverse events such as erythema, pain, swelling at the administration site, and fever, which usually resolve spontaneously without treatment. Serious adverse events related to the PVRV vaccine are rare, with an estimated incidence of 1 per 100,000 people.

Because of its proven safety record, this vaccine can be reasonably administered to healthy individuals. The established safety profile justifies our undertaking a non-inferiority trial in healthy individuals. However, our skilled staff will administer the vaccines properly while maintaining safety and asepsis to minimize any complications. We will conduct a follow-up assessment six months after the final vaccination to determine if any long-term adverse events have occurred and provide proper treatment if needed.

Vaccine Potency The quantifiable biological activity elicited by a vaccine antigen is known as its potency. According to the WHO, the potency of rabies vaccines should be 2.5 IU/intramuscular dose to elicit an adequate immune response once administered. 1 ml inj. Rabivax IM contains 2.5 IU of rabies antigen as per the potency recommended by WHO. On the other hand, the intradermal rabies vaccine regimen only requires a dose of 0.2 ml (0.1 ml in each arm), which corresponds to a potency of ≥0.5 IU/dose. Several studies showed a potency range of 0.22-2.32 IU/intradermal dose. Since the intradermal regimen requires multiple site administration and fractional dosing due to the abundance of antigen-presenting cells in the dermis, this antigen level in the vaccines is sufficient to produce immunogenicity similar to the levels of the IM regimen.

Appropriate Dosing According to the WHO guidelines, the intramuscular rabies vaccine regimen is given at a dose of 1 ml, while the intradermal regimen is given at a dose of 0.2 ml (0.1 ml in each arm). We will adhere to the guidelines since administration of 0.1 ml per intradermal site is considered appropriate for practical reasons and produces similar seroprotection levels. We will also administer 1 ml inj. Rabivax IM to the reference group per the recommended dosing schedule. As the WHO has already established and standardized the doses for both intradermal and intramuscular administration, we will not include an assessment of dose responses.

Appropriate Vaccine Schedule The dosing schedule for both intradermal and intramuscular rabies vaccine regimens has been included in the national guidelines. We will follow the 2-dose regimen for both vaccines. In the test group, 0.1 ml Inj. Rabivax will be administered intradermally on both the deltoid regions on days 0 and 7. We will administer 1 ml inj. Rabivax (2.5 IU/ml) vaccine intramuscularly on the deltoid region of one arm on days 0 and 7 in the reference group according to the instructions in the national guidelines.

Rationale Rationale of the non-inferiority trial According to the DGDA's regulatory requirements, a previously licensed and approved drug product requires additional approval to be marketed for administration via an alternate route. Therefore, a clinical trial comparing the non-inferiority of the intradermally administered rabies vaccine by Popular Pharmaceuticals PLC. to the intramuscularly administered rabies vaccine in terms of immunogenicity and safety can provide the foundation and evidence for its use in the Bangladeshi population.

Rationale of the age group The purified Vero cell vaccine for rabies has been proven to be remarkably safe and well-tolerated in children of all ages. This vaccine is already in use for people of all ages in Bangladesh, according to the National Guideline for Animal Bite Management. Therefore, we will assess the non-inferiority of the intradermal vaccine in terms of safety and immunogenicity across all age groups to strengthen the evidence generated by the trial, which is required for the vaccine's marketing authorization by the DGDA.

Rationale of the follow-up schedule We will conduct follow-up visits with the participants on days 21, 35, and 187. Since the RVNA level following vaccination peaks at 2-4 weeks, the first two follow-up visits will allow us to analyze the accurate seroconversion rate in the participants. We will perform a final follow-up for safety assessment on day 365 to assess the occurrence of any adverse effects that may manifest over the long term.

Suitability of the vaccine for the National Programme We will conduct this study at the Infectious Disease and Tropical Medicine Department (Surya Kanta Hospital), Mymensingh Medical College Hospital, Mymensingh. Since the National Guideline for Animal Bite Management in Bangladesh recommends the use of intradermal rabies vaccines for the management of rabies, it is likely that the study vaccine will be suitable for use by the National Programme.

Rationale for Pre-Exposure Prophylaxis Assessment This will be a non-inferiority trial evaluating the safety and immunogenicity of the intradermal rabies vaccine regimen, for which a licensed intramuscular regimen is already available. Therefore, we are exclusively assessing the pre-exposure prophylactic dosing of the rabies vaccine across both administration routes.

Benefits of the Participant Following Pre-exposure Vaccination Once the participants complete the PrEP regimen, routine booster doses will not be necessary for the general population. If an individual's RFFIT antibody titer remains ≥ 0.5 IU/mL (the minimum set by ACIP), they will be considered pre-immunized for any future rabies exposures. For any future exposures, only two doses of rabies vaccine would be needed for post-exposure prophylaxis, administered on days 0 and 7.

Justification for the exclusion of anamnestic response assessment:

Re-exposure to an antigen triggers a rapid, strong immune response known as an anamnestic response. As a part of this study, we are exclusively focusing on the safety and immunogenicity profile of the intradermal vaccine regimen. As the anamnestic response falls outside the parameters of our study objectives, we will not be investigating it.

Study Population and Sample Size:

We will recruit participants through community outreach and local advertisements. Interested individuals will be invited to the study site for an initial screening assessment. Before screening, potential participants will provide informed consent for the screening procedures. We will conduct a thorough assessment based on the established selection criteria. We will invite individuals meeting all eligibility criteria to participate in the study. Prior to enrollment, we will comprehensively explain the purpose, procedures, potential risks, and benefits of the study. We will provide ample opportunity for the participants to ask questions. We will enroll healthy individuals in the study following informed written consent. Each participant will be provided with a unique subject number that will be used for the identification of laboratory samples and all related documents throughout the study period. If a participant fails to qualify following the screening process, his/her subject number will not be allocated to another individual. Participants not satisfying the inclusion or exclusion criteria during the screening period will be considered screen failures. Data regarding the screen failures will be recorded in the source documents.

Study Design:

Non-inferiority of the intradermal regimen compared to the intramuscular regimen will be concluded if the lower bound of the two-sided 95% confidence interval for the difference in proportions (intradermal minus intramuscular) is greater than -5%. This non-inferiority margin of 5% has been chosen based on clinical considerations and regulatory guidance, as it represents a clinically acceptable difference in seroconversion rates between the two administration routes.

Screening and enrolment of the participants (-7 days):

To recruit healthy participants, we will utilize a combined local advertising and community outreach approach, including newspaper ads, cable TV broadcasts, leaflet distribution, and targeted university student outreach through campus-based information dissemination. This combination of advertising and outreach methods aims to maximize our reach and attract a diverse pool of eligible participants. Upon arrival at the study site, we will provide a comprehensive overview of the nature, purpose, benefits, and potential risks of the study to the interested individuals. After obtaining informed consent for the screening procedure, we will subject the participants to a thorough assessment using several inclusion and exclusion criteria. Upon successful completion of the eligibility assessment and confirmation by the study team, participants will be invited to enroll in the study. We will thoroughly explain the nature and purpose of our study. Additionally, we will inform them of the potential benefits and harms of administering the study vaccines. As per the Regulatory Authority in Bangladesh, free medical management and financial compensation will be provided to participants in case of study-related injury/death. They will be encouraged to ask questions regarding the study, and ample time will be provided to make informed decisions. After obtaining informed written consent, the investigator will keep the original, signed consent form with the study file. A copy of the signed informed consent form (ICF) will be provided to the subjects.

This single-period study will have a screening period of 7 days before the randomization process. Screening details will be documented in the screening log and recorded in the Site Master File. Participants will undergo a meticulous screening process by the research physician based on the following selection criteria.

Participant withdrawal:

Participants will be withdrawn/discontinued at any time during the study period on the occurrence of any of the following conditions-

1. The participant is no longer willing to participate in the study
2. If there is a protocol violation while enrolling the participant
3. Participant who has an adverse reaction to the study vaccine that threatens his/her well-being
4. Occurrence of any severe adverse event (SAE) or any symptoms or signs of extravasation as judged by the investigator
5. If the subject requires any concomitant vaccination for rabies or any other disease within the study period
6. Termination of study by sponsor
7. Investigator's discretion (for safety reasons).

Adverse events (AE)/Serious adverse events (SAE):

When a participant withdraws from participation during the study period, the investigator should document the reason clearly in the medical record and complete the designated page on the Case Report Form (CRF) describing the terms of discontinuation. Appropriate assessment must be ensured during all the visits.

During screening (Day -7), participants will undergo informed consent, eligibility assessment, demographic and medical history review, physical and systemic examination, vital signs measurement, ECG, pregnancy and infectious disease testing, laboratory investigations, and medication review. All medications taken 1 month before screening will be recorded at the screening visit. Following screening and enrollment, a unique identification number will be assigned to each subject, and their details (age, sex, weight, etc.) will be recorded in a corresponding file.

Following screening, enrolment, and assignment of treatment arms, subjects will be admitted on an outpatient basis and kept in the study ward during the vaccine administration period. General and systemic examinations will be performed before the vaccination, and vital signs will be assessed. Venous blood samples (10 mL) will be withdrawn within 5 minutes before vaccination on Day 0 to confirm a steady-state condition. Due to the brief seven-day period between screening and Day 0, we will rely on the screening blood test results (CBC, RBS, creatinine, SGPT, AST, and electrolytes) for efficiency and minimization of participant burden. This comprehensive baseline assessment will ensure the safety and validity of the trial.

The vaccines will be administered on Days 0 and 7 according to the pre-exposure prophylaxis (PrEP) regimen of the National Animal Bite Management Guideline. Proper aseptic measures will be maintained during vaccination, and expert personnel will administer the assigned vaccines. The participants will be observed for 30 minutes afterward, and any AE or SAE will be methodically recorded in the subject file.

Follow-up visits (Days 21 and 35):

Blood samples will again be collected on Days 21 and 35 to assess Rabies Virus Neutralizing Antibody (RVNA) in serum. According to the Advisory Committee on Immunization Practices guidelines, an RVNA level ≥ 0.5 IU/mL demonstrates an adequate response to vaccination (39). We will evaluate various blood parameters (CBC, SGPT, serum creatinine, serum electrolytes, AST) on day 21 and the RVNA level on days 21 and 35 to determine the safety and immunogenicity of the new vaccine regimen. Additionally, we will ensure that the participants do not take any concomitant medications during the study. The study physician will perform general and systemic examinations on Days 21 and 35, when AEs, SAEs, and vital signs will be assessed.

End of the study visit (Day 187):

On this visit, a total of 15 mL blood samples from each participant will be obtained for safety investigations and RVNA level assessment. We will record the vital signs and perform general and systemic examinations.

Concomitant medications will be checked for, and adverse events will be recorded. ECG recording will be performed to rule out any abnormality. After this thorough assessment, participants will be discharged from the hospital.

Blood for safety assessments at screening and the end of the study will be 15 mL. Total blood loss during the study will be 55 mL. Additional blood samples may be collected to ensure the safety of the participants during the study duration, as per the investigator's discretion.

Withdrawal Visit:

We will withdraw the participant from the study prematurely if he/she fulfill any of the withdrawal criteria specified in section II. The procedures to be performed on withdrawal include a general & systemic examination, vital signs assessment, clinical safety laboratory tests, and ECG. Furthermore, an AE assessment will be done. Details of concomitant medications will also be recorded.

Investigational Product Accountability:

The study vaccines, produced as a single lot, will be provided to the investigators by Popular Pharmaceuticals PLC. This medication must be stored securely in a locked, restricted-access area at the investigator's site and dispensed only to eligible participants under the investigator's or delegate's supervision. The vaccines must be stored according to the label's specified conditions. The investigator will document receipt of the vaccines. Dispensing and returns of study vaccines to trial participants will be recorded in IP logs provided by Popular Pharmaceuticals PLC. At study completion, the investigator will either retain all used, unused, defective, and reserved vaccines at the site or ship it to the third party, documenting this action. The investigator or a staff member must maintain accurate records of all study vaccine receipts and distribution using Drug Accountability Forms, which must be available for inspection.

Packaging and Labelling of Investigational Product Popular Pharmaceuticals PLC., Bangladesh, will supply study vaccines and provide them to the investigators. The vaccines will be packaged and labelled according to applicable regulations, including "For clinical trial use only" and, at a minimum, the active ingredient's name, participant number, study number, dosage form, directions for use, storage instructions, quantity, expiry date, batch number, and the sponsor and manufacturer's name and address. The investigational product will also be labelled per applicable study regulations. Study vaccines must be stored securely at the site, following protocol-specified conditions. Vaccine use will be thoroughly documented throughout the study. Unused vaccines and retention samples will be stored at the site or transferred to the manufacturers.

Method of Assigning Participants to Treatment Sequence:

This open-label study will use a 1:1 randomization (T/R) scheme to determine each participant's regimen. After a participant meets all eligibility criteria, provides informed consent, and is randomized, they will receive their assigned treatment. Participant numbers will remain consistent throughout the study, and participants may only participate once. Discontinued participants cannot be re-enrolled. If a participant withdraws consent after randomization or does not receive treatment for some reason, their assigned randomization number will not be reused.

Laboratory functions:

RVNA assessment:

We considered multiple time points to assess short and long-term antibody persistence. After discussion with the regulatory authority and considering the feasibility of the project, we decided to fix 14 and 28 days post-vaccination follow-up as short-term and 180 days post-vaccination as long-term follow-up timelines to assess the primary endpoint using the percentage of subjects in each group with a titre of IgG antibodies above the protective limits (≥ 0.5 IU/ml). Blood samples will be collected via an indwelling cannula in the antecubital vein. Post-dose samples will be collected within a scheduled time 3 days after vaccination, with the collection's end time recorded to the nearest minute. A +/- 30-minute window is allowed for post-dose sample collection. Every effort will be made to collect samples on time, and the actual collection time will be used in data analysis. If blood sample collection coincides with other study events (vitals), the following sequence will be followed: blood sample collection followed by vitals. RVNAs will be measured in serum samples using the RFFIT method as published in the WHO and OIE manuals. Briefly, 100 μL of each serum sample (in duplicate) will be serially diluted in 10% FBS-supplemented EMEM and loaded into 8-well Lab-Tek chamber slides. Then, 100 μL of the challenge virus (50TCID50) will be added. The slides will be incubated at 37 °C for 90 minutes, followed by the addition of 200 μL of a suspension of 5 × 10^5 BHK-21 C13 cells in 10% FBS-supplemented EMEM per well. They will then be placed in a 2-5% CO2 incubator at 37 °C for 24 hours. After incubation, the slides will be washed, fixed in 80% cold acetone, dried, and stained with FITC-conjugated anti-rabies antibody. Twenty fields per well will be examined under 100× magnification using a fluorescence microscope for rabies virus presence. RVNA titers will be calculated using the Reed-Muench method. Each test will include international standard rabies immunoglobulin (WHO SRIG), internal RVNA standards, and naïve serum as controls. SRIG will also serve as a calibrator for calculating sample IU/mL values.

ELISA:

We will further perform ELISA (Enzyme-Linked Immunosorbent Assay) to detect rabies antibodies in serum or plasma by utilizing rabies antigen coated onto a microplate. If antibodies are present, they will bind to the antigen and be subsequently detected using an enzyme-labeled secondary antibody. A substrate will then be added, producing a color change that correlates with the presence and concentration of rabies antibodies, which will be measured using a microplate reader. The process will involve several key steps: antigen coating, blocking of unbound sites, incubation with test and control samples, addition of the enzyme-labeled secondary antibody, substrate reaction, and absorbance measurement. Proper validation, inclusion of positive and negative controls, optimized dilutions, and thorough washing are crucial for accurate results. Biosafety precautions will be strictly followed when handling rabies antigens and samples. The procedure will be carried out as per the Standard Operating Procedure (SOP) of our collaborative organization.

Adverse Events (AE) Definition and Reporting:

An adverse event will be defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. It can, therefore, be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational treatment, whether considered related to the investigational treatment. The definition of an AE includes worsening (in severity and frequency) of pre-existing conditions/abnormalities ("Medical history") before the first Investigational Medicinal Product (IMP) administration and abnormalities of procedures (i.e., ECG, X-ray) or laboratory results, which are assessed as "clinically significant."

Serious Adverse Event (SAE):

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: Death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity, or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.

Adverse Event reporting period:

All adverse events (AEs) occurring within the specified reporting period must be reported to the DSMB. For non-serious AEs, reporting begins with the first dose of trial medication and continues until the checkout visit. Additionally, any non-serious AEs related to study procedures must be reported during the screening period (from informed consent signature). All serious adverse events (SAEs) must be reported from the time of informed consent signature until the end of the subject's trial participation.

Adverse event follow-up:

All adverse events (AEs) should be monitored until they resolve, are deemed chronic or stable by the investigator, or the subject's trial participation ends (i.e., until their final report is complete). Furthermore, all serious AEs and non-serious AEs considered possibly related to the investigational drug must be followed even after the subject's trial participation concludes. These events should be monitored until they resolve or are assessed as chronic or stable. The resolution of these events must be documented on the CRF and SAE forms.

Data Analysis:

A data entry program will be prepared using Microsoft Access. Data entry will be computerized and double-entered, followed by data quality control measures, including range and consistency checks. Discrepancies will be resolved by comparing the entered data with the original case report forms. Finally, all the data will be merged into a single database for statistical analysis using STATA version 17.

Data Safety Monitoring Plan:

Participant confidentiality will be rigorously protected and reported to the DSMB. If the interim analysis data cause the initial hypothesis/specific aims to be substantially reconsidered, we will seek guidance from the DSMB for further approaches to be taken to complete the study. The final meeting will be held at the end of the study. In addition to that, any SAE will be reported to the DSMB immediately, and the study will be stopped until further direction by the DSMB is received. All AEs will be recorded in the participant information form. Data Monitoring will be unblinded.

Collaborative Arrangements:

We will collaborate with the Institut für molekulare Virologie und Zellbiologie, which is a WHO reference laboratory in Germany. We will ship the samples to our collaborator, who will help us with the RFFIT and ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged >4 years
* Able to comply with the research process and provide informed consent
* Able to attend all the scheduled visits and comply with the trial procedures
* Medical history and clinical examination demonstrating that the subject is healthy
* Women willing to follow any method of contraception throughout the duration of the study.

Exclusion Criteria:

* Subjects participating in other clinical trials in the 4 weeks preceding the first trial vaccination dose
* Subjects with a history of previous rabies vaccination (either pre- or post-exposure prophylaxis)
* Subjects with a history of receiving Rabies immunoglobulin (Ig (human/equine) prior to the study
* Subjects with a fever (≥37.2°C) or any moderate or severe acute illnesses or active infections on the day of vaccination
* History of systemic hypersensitivity to any component included in the vaccine or a history of adverse events as a reaction to previous experimental vaccine studies
* History of receiving any immunoglobulin, blood, or blood-based product in the last 3 months or planning to donate blood in the following 3 months, which may interfere with the immune response
* Screened as positive for HBsAg, Anti-HCV, and anti-HIV
* Subjects receiving any vaccine at least 4 weeks prior to enrolment or expected to receive any vaccine 4 weeks after the administration of the trial vaccine.
* Lactating women or pregnant women as detected by the urine hCG strip test.
* History of alcohol or any substance abuse (benzodiazepines, methamphetamines, opioids, cannabinoids, cocaine, barbiturates) within 1 year
* Subjects with congenital or acquired immunodeficiency or subjected to short- or long-term corticosteroid or immunosuppressive therapy
* Thrombocytopenia, bleeding disorders, or anticoagulants used during the 3 weeks prior to trial vaccination to avoid intramuscular haemorrhage
* Any major psychiatric disorder such as schizophrenia, major depressive disorder, severe anxiety disorder, etc.
* History of cardiac arrhythmias, such as bradycardia, tachycardia, supraventricular tachycardia (SVT), ventricular tachycardia (VT), ventricular fibrillation (VF), atrial fibrillation (AF), etc., as assessed by the electrocardiogram report
* History of renal insufficiency or dialysis
* Any immunosuppressive disorder, such as cancers, multiple myeloma (MM), various autoimmune diseases, etc.
* Participants with clinically significant or abnormal laboratory parameters (serum creatinine, SGPT, AST, serum electrolytes) in the opinion of the investigator.
* Any condition that presents an unacceptable risk of injury, as assessed by the site investigator
* Subjects planning to have surgery in the 3 months preceding the completion of the project
* Subjects concurrently using anti-malarial drugs
* Any condition that, in the researcher's opinion, would jeopardize the safety or rights of the subject or prevent the subject from completing the procedures of the study protocol
* Subjects exposed to any rabid animal bite in the 4 weeks preceding the commencement of the study.
* Subjects with Type I or Type II Diabetes, as assessed by Random Blood Sugar level.
* All research facility staff directly participating in this study, including their immediate family and relatives.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate | 14 days, 28 days, and 180 days following the completion of vaccination doses
  Rabies Virus Neutralizing Antibody: ≥ 0.5 IU/mL

SECONDARY OUTCOMES:
Number of participants with treatment-related serious adverse events as assessed by CTCAE v5.0 | Participants will be followed up 14 days, 28 days, and 180 days following the completion of vaccination doses. They will also contact the research team for self-reporting of adverse events.
  Zero serious adverse events reported by the participants by the end of the study will be considered as a safety measure.
Number of participants with post-vaccination laboratory abnormalities | The number of participants with post-vaccination laboratory values will be assessed on day 21 and day 187 of the study.
  Number of participants with clinical laboratory values outside the following reference ranges will be zero:
  i. Haemoglobin: 13.5 to 17.5 g/dL in adult males, 12 to 16 g/dL in adult females, 12.5 to 16.1 g/dL in male children of 10-17 years, 12 to 15 g/dL in female children of 10-17 years, 11.5 to 14.5 g/dL in children aged 5-9 years.
  ii. Red blood cell count: 4.3 to 5.7x10^8/mm3 in adults, 3.5 to 4.7x10^8/mm3 in children aged 10-17 years, and 3.3 to 4.3x10^8/mm3 in children aged 5-9 years.
  iii. Platelet count: 150 to 400 x 103/mm3 iv. Total white blood cell count: 4.5 to 11 x 103/mm3 a. Neutrophils: 57%-67% b. Lymphocytes: 23%-33% c. Monocytes: 3%-7% d. Eosinophils: 1%-3% e. Basophils: 0%-1% v. Serum Electrolytes -
  1. Na+: 135-145 mmol/L
  2. K+: 3.5-5.3 mmol/L
  3. Mg2+: 0.6-1.1 mEq/L
  4. Cl-: 98-108 mmol/L vi. Random Blood Sugar: <200 mg/dL vii. Renal Function test: creatinine: 0.6-1.3 mg/dL viii. Liver Function Test -
  a. SGPT: 3 to 48 U/L b. Aspartate Aminotransferase (AST): 0 to 55 U/L
Number of participants with post-vaccination abnormalities in vital signs | Vital signs will be evaluated on the day of check-in (day 0), day 7, and during post-vaccination follow-up (day 21, 35, and 187); 30 minutes before dosing on vaccination days
  There will be no clinically significant deviation from these normal ranges in all participants:
  i. Oral temperature: 97°F to 99°F. ii. Respiratory rate: 15 to 25 breaths/min in children aged 5 to 9, 15 to 20 breaths/min in children aged 10 to 17, and 12 to 20 in individuals aged 18 years and above.
  iii. Blood pressure (BP): 120 to 129 systolic BP and 70-90 Diastolic BP. iv. Pulse rate: 60 to 100 beats per min.
Number of participants with post-vaccination abnormalities found in physical examination | General and systematic examination will be conducted on check-in (Day 0), day 7, and during post-vaccination follow-up (Days 21, 35, and 187) and
  A complete general and systemic examination will be conducted by a physician including (at a minimum) a thorough examination of the following:
  General and Systemic examination includes the Head, Neck, Eyes, Ears, Nose, Throat, skin and appendages, Renal, Cardiovascular, Pulmonary, Urology, Reproductive, Endocrine, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shomik Maruf, MSc, Principal Investigator — International Center for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Infectious Disease and Tropical Medicine Department (Surya Kanta Hospital), Mymensingh Medical College Hospital, Mymensingh, Mymensingh, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive personal and clinical information that could compromise participant confidentiality. Furthermore, there is no specific plan or ethical approval in place for secondary data sharing beyond the current study objectives. Only aggregated, de-identified results will be disseminated through publications and presentations.

REFERENCES:
- [Background] World Health Organization. WHO guidelines on non-clinical evaluation of vaccines, Annex 1, TRS No 927
- [Background] World Health Organization. WHO Expert Consultation on Rabies: WHO TRS N°1012. 2018
- [Background] Guideline for Animal Bite Management in Bangladesh 2021